CLINICAL TRIAL: NCT00989482
Title: Improving Antibiotic Prescribing Practices in Mexican Primary Care Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Ralph Gonzales, University of California, San Francisco
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Fulbright-Gonzales
Record Dates: First submitted 2009-07-24; First posted 2009-10-05 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Acute Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Computer Kiosk Eduction (Experimental)
  Interventions: Behavioral: Computer kiosk Education

INTERVENTIONS:
Behavioral: Computer kiosk Education — computerized patient education; guidelines for physicians

SUMMARY:
The purpose of this study is to improve antibiotic prescribing practices of Mexican primary care physicians for patients seeking care for acute respiratory tract infections (ARIs). The investigators will employ a combination of qualitative and quantitative methods to develop and evaluate a patient education and physician decision-support intervention.

Hypothesis 1: The investigators will identify barriers and facilitators of appropriate antibiotic use for ARIs that can be addressed through patient education and physician decision-support.

Hypothesis 2: The proportion of patients who report desire for antibiotics as a "very important" reason for seeking care will decrease from 50% to 30% following exposure to the educational intervention; and 90% (95% confidence interval: 80% to 100%) of patients will report that they trust the information provided by the computer.

Hypothesis 3: Antibiotic prescribing for adults with uncomplicated acute bronchitis will decrease from 80 percent to 40 percent following the introduction of a real-time clinical decision support tool.

ELIGIBILITY:
Inclusion Criteria:

* adults age 18 years or greater

Exclusion Criteria:

* mental disability; severe illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 847 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
antibiotic prescription rate | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- IMSS Family Practice Clinic #1, Cuernavaca, Morelos, Mexico